CLINICAL TRIAL: NCT05801094
Title: A Phase I Clinical Study to Evaluate Safety、 Tolerability, and Pharmacokinetics of QL1604 for the Treatment of Advanced Solid Tumors - A Phase Ic Preliminary Efficacy Expansion Study
Brief Title: A Phase I Study of QL1604 for Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QL1604-002
Record Dates: First submitted 2023-03-24; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QL1604 (Experimental)
  Interventions: Drug: QL1604

INTERVENTIONS:
Drug: QL1604 — QL1604 3 mg/kg Q3W

SUMMARY:
In this study, patients with advance solid tumors will be treated with QL1604 monotherapy.

ELIGIBILITY:
Key Inclusion Criteria:

* 18-75 years;
* At least one measureable lesion as defined per RECIST Version (v) 1.1
* Histologically or cytologically confirmed、failed to standard therapy or lack standard therapy(except immunotherapy) advanced solid tumors; for cervical cancer, only squamous carcinoma、adenocarcinoma、adenosquamous carcinoma could be enrolled； hepatocellular carcinoma could be enrolled by clinical diagnosis
* Adequate important organ function

Key Exclusion Criteria:

* Active autoimmune disease orautoimmune disease history
* Meningeal metastasis,or brain metastasis( except asymptomatic brain metastasis, or symptomatic brain metastasis but stable for more than 4 weeks after treatment, and have stopped systemic hormone treatment (prednisone of > 10 mg/day or equivalent hormone) for more than 2 weeks)
* Known hypersensitivity to protein macromolecules, and/or any of QL1604 excipients
* Radiotherapy, chemotherapy, hormone therapy, surgery, targeted therapy within 4 weeks prior to study drug (for micromolecule targeted therapy, within 2 weeks)
* Active hepaititis B or C infection
* Both HBsAg and anti-HCV Ab positive

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2023-04-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | up to 2 years
  ORR is defined the percentage of the participants who have achieved complete response (CR) or partial response (PR) using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 after the initiation of study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Weijian Guo, PhD, Study Chair — Fudan University; Jianping Xiong, PhD, Study Chair — The First Affliated Hospital of Nanchang University
Locations (2):
- China (2):
  - The First Affliated Hospital of Nanchang University, Nanchang
  - Fudan University Shanghai Cancer Center, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xiong J, Ouyang W, Yang M, Gao Z, Zhou H, Lou H, Guo Y, Xu Z, Zheng L, Liu Y, Wang Z, Sun P, Niyazi H, Wang J, Chen Y, Zhang B, Li L, Kang X, Guo W. Efficacy and Safety of Iparomlimab, an Anti-PD-1 Antibody, in Patients with Advanced Solid Tumors: A Phase 1c Study. Adv Ther. 2024 Nov;41(11):4153-4171. doi: 10.1007/s12325-024-02981-z. Epub 2024 Sep 14. PMID 39276185